CLINICAL TRIAL: NCT04459832
Title: Optimal Time of Hamstring Stretch in Elderly
Brief Title: Optimal Duration of Stretching of the Hamstring Muscle Group in Elderly: A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shimaa Taha Abu El Kasem, Lecturer of Physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A Randomized Controlled Trial
Record Dates: First submitted 2020-06-25; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Stretch
Keywords: Stretching; Randomized controlled trial; Hamstring

STUDY DESIGN:
Intervention Model Description: randomized controlled trial study 100 participants will be recruited to participate in the study after assigning a conset form, participants will be divided into 4 group ,one control which will not receive stretch of hamstring and 3 experimental groups will recive different duration for hamstring stretch 15,30,60 and DSSEP will be measured as the primary outcome and knee ROM will be measured as a secondary outcomes in order to identify the optimal duration of hamstring stretch
Who Masked: Participant
Masking Description: The assessor, who took the measurements for both the intervention and control groups, was blinded to the subject's group, while the treating therapist was not blinded to the treatment intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 15 second stretch (Experimental): Stretching of the hamstring muscles was performed by the primary researcher for 15 seconds. A straight-leg-raising technique was used for this stretch because we believe that it is commonly used in the clinical setting for elderly people. All subjects were supine lying as flat as possible
  Interventions: Procedure: stretch hamstring
- 30 second stretch (Experimental): Stretching of the hamstring muscles was performed by the primary researcher for 30 seconds. A straight-leg-raising technique was used for this stretch because we believe that it is commonly used in the clinical setting for elderly people. All subjects were supine lying as flat as possible
  Interventions: Procedure: stretch hamstring
- 60 second stretch (Experimental): Stretching of the hamstring muscles was performed by the primary researcher for 60 seconds. A straight-leg-raising technique was used for this stretch because we believe that it is commonly used in the clinical setting for elderly people. All subjects were supine lying as flat as possible
  Interventions: Procedure: stretch hamstring
- control (Sham Comparator): The control group followed the same procedures except that no stretching force was applied at the end
  Interventions: Procedure: stretch hamstring

INTERVENTIONS:
Procedure: stretch hamstring — Stretching of the hamstring muscles was performed by the primary researcher. A straight-leg-raising technique was used for this stretch because we believe that it is commonly used in the clinical setting for elderly people. All subjects were supine lying as flat as possible

SUMMARY:
identification of optimal duration for hamstring muscle stretch by using 3 different time of stretch 15,30,60 seconds .100 subjects will be participated in this study divided into 4 group one control and 3 experimental groups according to stretch time.

DETAILED DESCRIPTION:
Abstract:

OBJECTIVE: To explore the effect of variable stretching intervals on neural function and ROM.

DESIGN: Randomized controlled trial Participants: In this trial, 100 participants will participate in the study diagnosed with tight hamstring muscles (defined as the inability to extend the knee to less than 20° of knee flexion) were randomly assigned to the control group or one of the 3 intervention groups Interventions: The three experimental groups will stretched 5 times per week for 4 weeks for 15, 30, and 60 seconds, respectively the control group did not stretch Main Outcome Measures: The neurophysiological outcome measures included peak to peak somatosensory evoked potential for dermatomes L3,L4,L5, and S1. Secondary outcome measures included knee ROM. All outcome measures will be assessed immediately after the treatment session and 24 hours after the treatment session.

ELIGIBILITY:
Inclusion Criteria:

* Subjects had to demonstrate "tight" hamstring muscles, defined as inability to extend the knee to less than 20 degrees of knee flexion with the femur held at 90 degrees of hip flexion while the person was positioned supine. Subjects were also screened to rule out knee joint flexion contractures by checking knee extension ROM, while they were lying in a prone position

Exclusion Criteria:

* Using of medical aids, and suffering from any neurological or cognitive impairment, limiting cardio-respiratory conditions, or had undergone recent surgery (within the past 12 months). Having any hip or knee replacements or any history of pathology in the low back, hips, or knees for the 3 months prior to the study

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Neurophysiological findings. | Assessments of the change of DSSEPs from baseline to immediatly after session and at 24 hour after session
  Neurophysiological findings included peak to peak somatosensory evoked potentials (DSSEPs) for L3,L4,L5,S1 dermatomes.

SECONDARY OUTCOMES:
ROM | Assessments of the change of Knee ROM from baseline to immediatly after session and at 24 hour after session
  Each subject was then measured for knee extension ROM on both lower extremities

IPD SHARING:
Plan to Share IPD: No